CLINICAL TRIAL: NCT04985370
Title: Pain Neuroscience Education Plus Exercise Versus Exercise Alone in the Management of Chronic Rotator Cuff Tendinopathy: a Randomized Controlled Trial
Brief Title: PNE Plus Exercise Versus Exercise for Chronic Rotator Cuff Tendinopathy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic issues
Sponsor: Ruben Fernandez Matias (Other)
Responsible Party: Sponsor-Investigator, Ruben Fernandez Matias, Clinical Professor, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/58
Record Dates: First submitted 2021-07-20; First posted 2021-08-02 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Rotator Cuff Tendinosis
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers involved in recording outcome measures will not be aware of treatment allocation. Patients will be encouraged to not tell the evaluators about the received treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education plus exercise (Experimental): Three sessions of pain neuroscience education plus exercise.
  Interventions: Other: Pain neuroscience education; Other: Exercise
- Exercise alone (Active Comparator): Exercise alone without pain neuroscience education.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Pain neuroscience education — Three sessions of pain neuroscience education based on explaining patients: characteristics of acute versus chronic pain, function of acute pain, how acute pain is originated within the nervous system, how acute pain progress to chronic pain, and factors that contribute to central sensitization (e.g., emotions, stress, disease and pain beliefs, behaviors regarding pain...). All the explanations will be conducted using easy-understandable examples and metaphors.
  Arms: Pain neuroscience education plus exercise
Other: Exercise — Progressive resistance exercise program based on isometric, concentric, eccentric, and pliometric contractions.

SUMMARY:
The aim of this randomized controlled trial is to evaluate the combined effects of pain neuroscience education plus exercise to exercise alone in the management of patients with chronic rotator cuff tendinopathy regarding pain, function, strength, kinesiophobia, and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain due to rotator cuff tendinopathy lasting more than 6 months.
* Internal Rotation Resisted Strength Test positive.
* Test Item Cluster (Hawkins-Kennedy, painful arc, and infraspinatus test) positive.

Exclusion Criteria:

* History of: tumors, metastasis, osteoporosis, shoulder fractures, shoulder luxation and/or instability, previous shoulder surgery, cervical radiculopathy, full-thickness rotator cuff tears, glenohumeral joint degeneration, inflammatory arthropathy, acromioclavicular joint arthrosis, and rotator cuff calcifications.
* Being treated by other physical therapy or medical treatment for their shoulder pain at the time of recruitment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-07-25 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline, change from baseline at 4-week, and change from baseline at 12-week
  Pain intensity measured with numerical pain rating scale which ranges from 0 points (no pain) to 10 points (worst imaginable pain)

SECONDARY OUTCOMES:
Shoulder disability change | Baseline, change from baseline at 4-week, and change from baseline at 12-week
  Shoulder disability measured with Shoulder Pain and Disability Index (SPADI). SPADI ranges from 0% (no disability) to 100% (maximum degree of disability).
Kinesiophobia change | Baseline, change from baseline at 4-week, and change from baseline at 12-week
  Kinesiophobia measured with Tampa Scale for Kinesiophobia (TSK-11) which ranges from 0% (no kinesiophobia) to 100% (maximum degree of kinesiophobia).
Catastrophism change | Baseline, change from baseline at 4-week, and change from baseline at 12-week
  Catastrophism measured with Pain Catastrophizing Scale (PCS) which ranges from 0% (no catastrophism) to 100% (maximum degree of catastrophism).
Strength change | Baseline, change from baseline at 4-week, and change from baseline at 12-week
  Scaption strength at 90º of elevation measured with a hand-held dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Rubén Fernández-Matías, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No